CLINICAL TRIAL: NCT02907021
Title: A Phase I Clinical Study to Examine the Safety of Continued Treatment With Trastuzumab for Individuals With Overt Left Ventricular Dysfunction
Brief Title: Safety of Continuing CHemotherapy in Overt Left Ventricular Dysfunction Using Antibodies to HER-2
Acronym: SCHOLAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHOLAR-2016
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure; Breast Cancer
MeSH Terms: conditions — Heart Failure; Breast Neoplasms | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heart failure (Experimental): Treat the HER-2 positive breast cancer patients experiencing mild or moderate LV impairment by standard-of-care treatments for LV impairment using ACE-I and beta-blockers
  Interventions: Drug: standard-of-care treatments for LV impairment

INTERVENTIONS:
Drug: standard-of-care treatments for LV impairment — Treat patients with mild or moderate LV impairment by standard-of-care treatments for LV impairment using ACE-I and beta-blockers
  Other Names: ACE-I and beta-blockers

SUMMARY:
Trastuzumab is an important treatment for HER 2 positive breast cancer. But trastuzumab can cause injury to the heart, and this is one of the main reasons it cannot be administered as planned. Heart injury can often be successfully treated using cardiac medications. The aim of SCHOLAR is to evaluate whether it is safe to continue trastuzumab in individuals with mild or moderate cardiac injury, while treating them with appropriate cardiac medications. In this way the investigators hope to be able to optimise the delivery of a treatment to patients with breast cancer that has proven survival benefits, especially when administered for a full 12-month course.

DETAILED DESCRIPTION:
The SCHOLAR study design will be a modified phase I, non-randomized clinical study.

Initially a cohort of 5 participants will be enrolled. They will continue to receive trastuzumab. All participants in SCHOLAR will also be prescribed standard-of-care treatment for patients with LV systolic dysfunction, including the beta-blocker, carvedilol, and the ACE-I, ramipril, as tolerated, at the maximum doses tolerated, up to carvedilol 25mg BID and ramipril 10mg once daily. If at any time 1 or more of the first 5 participants develop cDLT, de-escalation will occur. De-escalation will involve a change in the eligibility criteria to exclude patients with LVEF <45% and patients with NYHA class II, III, or IV heart failure. A further 5 patients will then be recruited. If 2 or more of the second 5 participants develop cDLT after de-escalation, the intervention will be considered unsafe, and the study will be closed. If the intervention is considered safe either using the initial eligibility criteria or the de-escalated eligibility criteria, the study will be closed after 20 participants have been recruited. If at any time during the study >20% of participants develop cDLT, the intervention will be considered unsafe, and the study will be closed.

Patients will be seen by a cardiologist at the following time points (referenced from the baseline visit): baseline, 3 weeks ± 1 week, 6 weeks ± 1 week, 3 months ± 1 week, 6 months ± 1 week, 9 months ± 1 week, 12 month ± 1 week

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III HER-2 positive breast cancer
* Receiving adjuvant therapy with trastuzumab
* Provide informed consent
* Exhibit LV dysfunction as evidenced by either

  * LVEF between 40% and the lower limit for normal (i.e. <54% in women or < 52% in men18), or
  * LVEF within normal limits (i.e. ≥54% in women or ≥52% in men) and NYHA class II heart failure symptoms within the past year, or
  * A fall in LVEF of ≥15% from baseline

Exclusion Criteria:

Patients will not be eligible for SCHOLAR if they have any of the following:

* NYHA class III or IV heart failure
* Systolic blood pressure <90mmHg
* Current use of both ACE-I/angiotensin receptor blocker and beta-blocker
* Contra-indication to both ACE-I/angiotensin receptor blocker and beta-blocker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Safety outcomes | one year
  The primary safety outcome will be the development of cardiac dose-limiting toxicity (cDLT), defined as the occurrence of any of a)cardiovascular death, b)left ventricular ejection fraction (LVEF) <40% together with any heart failure symptoms, or c) LVEF <35%
Efficacy outcomes | one year
  The efficacy outcome will be the number of trastuzumab cycles completed after enrollment as a proportion of the originally planned number of trastuzumab cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Leong, PhD. MBBSm, Principal Investigator — Population Health Research Institute
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leong DP, Cosman T, Alhussein MM, Kumar Tyagi N, Karampatos S, Barron CC, Wright D, Tandon V, Magloire P, Joseph P, Conen D, Devereaux PJ, Ellis PM, Mukherjee SD, Dhesy-Thind S. Safety of Continuing Trastuzumab Despite Mild Cardiotoxicity: A Phase I Trial. JACC CardioOncol. 2019 Jul 17;1(1):1-10. doi: 10.1016/j.jaccao.2019.06.004. eCollection 2019 Sep. PMID 34396157